CLINICAL TRIAL: NCT03024905
Title: Enhancing All Community Health Workers on Maternal and Newborn Health: Rorya Tanzania
Brief Title: Project to Use Community Health Workers to Reduce Maternal Deaths
Acronym: EWH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: Ottawa Hospital Research Institute (Other); Shirati KMT Hospital (Unknown)
Responsible Party: Principal Investigator, Gail Webber, Associate Scientist, Bruyère Health Research Institute.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 108026
Record Dates: First submitted 2016-12-11; First posted 2017-01-19 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Maternal Mortality; Access to Health Care
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Division 1 (Experimental): The first division receives baseline data collection for 6 months then experiences interventions for the remainder of the trial.
  Interventions are behavioural and device:
  Behavioural: education about safety of delivery at a health facility, reminders to go for antenatal care, and a voucher for transport to the health facility at the time of delivery.
  Device: A birth kit with clean delivery supplies (soap, 2 pairs of gloves, cord clamps, surgical blade, and 600 mcg misoprostol for the woman to take immediately after the delivery to prevent postpartum hemorrhage).
  Interventions: Behavioral: Village meeting and travel vouchers; Device: Birth kit with misoprostol
- Division 2 (Experimental): The second division receives baseline data collection for 9 months then experiences interventions for the remainder of the trial.
  Interventions are behavioural and device:
  Behavioural: education about safety of delivery at a health facility, reminders to go for antenatal care, and a voucher for transport to the health facility at the time of delivery.
  Device: A birth kit with clean delivery supplies (soap, 2 pairs of gloves, cord clamps, surgical blade, and 600 mcg misoprostol for the woman to take immediately after the delivery to prevent postpartum hemorrhage).
  Interventions: Behavioral: Village meeting and travel vouchers; Device: Birth kit with misoprostol
- Division 3 (Experimental): The third division receives baseline data collection for 12 months then experiences interventions for the remainder of the trial.
  Interventions are behavioural and device:
  Behavioural: education about safety of delivery at a health facility, reminders to go for antenatal care, and a voucher for transport to the health facility at the time of delivery.
  Device: A birth kit with clean delivery supplies (soap, 2 pairs of gloves, cord clamps, surgical blade, and 600 mcg misoprostol for the woman to take immediately after the delivery to prevent postpartum hemorrhage).
  Interventions: Behavioral: Village meeting and travel vouchers; Device: Birth kit with misoprostol
- Division 4 (Experimental): The fourth division receives baseline data collection for 15 months then experiences interventions for the remainder of the trial.
  nterventions are behavioural and device: Behavioural: education about safety of delivery at a health facility, reminders to go for antenatal care, and a voucher for transport to the health facility at the time of delivery.
  Device: A birth kit with clean delivery supplies (soap, 2 pairs of gloves, cord clamps, surgical blade, and 600 mcg misoprostol for the woman to take immediately after the delivery to prevent postpartum hemorrhage).
  Interventions: Behavioral: Village meeting and travel vouchers; Device: Birth kit with misoprostol

INTERVENTIONS:
Behavioral: Village meeting and travel vouchers — The interventions are:
  1. Village meetings by community health workers to educate women and their families about safe birthing.
  2. Vouchers for free transport by motorcycle taxi drivers to access health facility at delivery.
Device: Birth kit with misoprostol — Provision of birth kit with clean delivery supplies (soap, 2 pairs of gloves, 2 cord clamps, surgical blade, and 600 mcg misoprostol for the woman to take immediately after the delivery to prevent postpartum hemorrhage).

SUMMARY:
The purpose of this trial is to establish if several interventions will help women in rural Tanzania access health care services during pregnancy and at the time of delivery. The interventions include education about the importance of attending antenatal care visits with nurses and facility deliveries, a voucher for transport to access the health facility at the time of delivery, and supplies to be used either at the health facility, or on route if the women does not make it to the health facility.

DETAILED DESCRIPTION:
In order to reduce the number of women dying in childbirth and to improve women's health in pregnancy, this trial is designed to assess if several interventions combined can increase the number of women delivering in health care facilities. The design of the study is "Multiple Baseline Design". Community health workers are trained to collect baseline data on women using mobile phones in one rural district in Tanzania. The district has four distinct divisions. After 6 months of baseline data in the district, one division will experience the interventions. The interventions are education about the importance of attending antenatal care visits with nurses and facility deliveries, a voucher for transport to access the health facility at the time of delivery, and birthing supplies to be used either at the health facility, or on route if the women does not make it to the health facility. The intervention will be begun in each of the other divisions in 3 month intervals (i.e. the second division starts to experience the interventions 3 months after the first, the third, 3 months after the second and the fourth 3 months after the third). The trial will continue for a total of 27 months including the baseline period.

ELIGIBILITY:
Inclusion Criteria:

1. Women must be pregnant.
2. Women must live in Rorya District, but not in Shirati Town.
3. Women must deliver in Rorya District .

Exclusion Criteria:

1. Women who live outside or deliver outside of Rorya District.
2. Women who deliver preterm, before they have exposure to all the interventions.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17000 (Estimated)
Dates: Start 2017-01-16 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Facility births | During baseline vs during intervention periods until end of study (2 years)
  Number of women attending health facilities for delivery

SECONDARY OUTCOMES:
Antenatal Care visits | During baseline vs during intervention until end of study (2 years)
  Number of times women attend health facility for antenatal visits
Postpartum visits | During baseline vs during intervention until end of study (2 years)
  Number of women attending health facility for postpartum visits
Use of transport intervention | During Intervention until end of study (2 years)
  Number of women using the free transport intervention
Use of birth kit | During Intervention until end of study (2 years)
  Number of women using the birth kit

CONTACTS AND LOCATIONS:
Overall Officials: Bwire Chirangi, MPH, Principal Investigator — Director of Shirati KMT Hospital; Gail C Webber, MD, PhD, Principal Investigator — Bruyère Health Research Institute.
Locations (1):
- Shirati District Hospital Research Office, Shirati, Rorya District, Mara, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Webber G, Chirangi B, Magatti N, Mallick R, Taljaard M. Improving health care facility birth rates in Rorya District, Tanzania: a multiple baseline trial. BMC Pregnancy Childbirth. 2022 Jan 27;22(1):74. doi: 10.1186/s12884-022-04408-5. PMID 35086508